CLINICAL TRIAL: NCT02288195
Title: Phase III Study of Neoadjuvant Chemotherapy With Capecitabine and Oxaliplatin Versus Chemoradiation for Locally Advanced Rectal Cancer Patients
Brief Title: CONVERT: Neoadjuvant Chemotherapy Alone Versus Preoperative Chemoradiation for Locally Advanced Rectal Cancer Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Shantou Central Hospital (Other); Liaoning Cancer Hospital & Institute (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Fujian Cancer Hospital (Other Government); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); First Affiliated Hospital of Chongqing Medical University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Guangdong Provincial People's Hospital (Other); Cancer Hospital of Guangxi Medical University (Other); Meizhou People's Hospital (Other); Henan Cancer Hospital (Other Government); Affiliated Cancer Hospital of Shantou University Medical College (Other); Hubei Cancer Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); Longyan City First Hospital (Other); Shengjing Hospital (Other); Zhejiang Cancer Hospital (Other); Jiangmen Central Hospital (Other); West China Hospital (Other); The Third Affiliated Hospital of Kunming Medical College. (Other)
Responsible Party: Principal Investigator, Pei-Rong Ding, Associate Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT02288195
Record Dates: First submitted 2014-02-24; First posted 2014-11-11 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Rectal Neoplasms
Keywords: Neoadjuvant Chemotherapy; Preoperative radiotherapy; Chemoradiotherapy; Capecitabine; Oxaliplatin
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Capecitabine; Radiation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chemotherapy (Experimental): Patients receive neoadjuvant chemotherapy comprising oxaliplatin 130mg/m² ivdrip over 2 hours on day 1,capecitabine 2000 mg/m² on days 1-14, treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.Patients without disease progression undergo low-anterior resection (LAR) with total mesorectal excision (TME) and 4 cycles of XELOX ( oxaliplatin 130mg/m² day 1，capecitabine 2000mg/m² days 1-14, repeated every 21 days). Patients with disease progression undergo chemoradiation as in group chemoradiotherapy before proceeding to LAR with TME.
  Interventions: Drug: Oxaliplatin; Drug: capecitabine
- Chemoradiotherapy (Experimental): Patients receive capecitabine 825 mg/m² twice daily concurrently with radiation therapy for 5 days per week. Patients also undergo intensity-modulated radiation therapy 5 days a week for approximately 5.5 weeks. Patients then undergo LAR with TME and 4 cycles of XELOX ( oxaliplatin 130mg/m² day 1，capecitabine 2000mg/m² days 1-14, repeated every 21 days) .
  Interventions: Drug: capecitabine; Radiation: Radiation

INTERVENTIONS:
Drug: Oxaliplatin — 130 mg/m² iv drip over 2 hours on day 1, repeated every 21 days.
  Other Names: Eloxatin
  Arms: Chemotherapy
Drug: capecitabine — 825 mg/m² twice daily administered orally and concurrently with radiation therapy for 5 days per week.
  1000 mg/m² po twice daily on days 1- 14 repeated every 21 days in Group A and adjuvant chemotherapy in Group B.
  Other Names: Xeloda
Radiation: Radiation — The total dosage was 46Gy consisted of 23 fractions of 2 Gy to clinical target volume without a boost dose and with the boost 4 Gy consisted of 2 fractions of 2 Gy to gross tumor volume by IMRT or 3D-CRT.
  Other Names: radiotherapy
  Arms: Chemoradiotherapy

SUMMARY:
Although neoadjuvant radiotherapy greatly decreases local recurrence in locally advanced rectal cancer patients undergoing surgery, it inevitably results in short-term and long-term toxicities. More importantly, it has not been confirmed that neoadjuvant radiotherapy could improve overall survival. The purpose of this study is to compare the effects of chemotherapy alone using a combination regimen known as XELOX (capecitabine and oxaliplatin ) and selective use of the standard treatment to the standard treatment of chemotherapy and radiation.

DETAILED DESCRIPTION:
This randomised, open-label, multicentre,phase 3 trial began in August, 2014, as an adjuvant trial comparing capecitabine-based neoadjuvant chemoradiotherapy with chemotherapy alone,in patients aged 18 years to 75 with clinical stage II-III locally advanced rectal cancer from six Chinese institutions.

Patients with local advanced rectal cancer (T2N+ or T3-4aNany,M0, CRM≥2mm, 12cm from the anus verge) were scheduled to Group A: receive neoadjuvant chemotherapy alone (4 cycles of XELOX: oxaliplatin 130mg/m2 day 1，capecitabine 2000mg/m2 days 1-14, repeated every 21 days) followed by radical surgery and 4 cycles of XELOX ( oxaliplatin 130mg/m2 day 1，capecitabine 2000mg/m2 days 1-14, repeated every 21 days) and Group B :chemoradiotherapy (50.4 Gy plus capecitabine 1650 mg/m² administered orally and concurrently with radiation therapy for 5 days per week.) followed by radical surgery and 6 cycles of XELOX ( oxaliplatin 130mg/m2 day 1，capecitabine 2000mg/m2 days 1-14, repeated every 21 days) The primary endpoint was 3-year local recurrence free survival; analyses were done based on all patients with post-randomization data.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Diagnosis of rectal adenocarcinoma
* Radiologically measurable or clinically evaluable disease
* Tumor location within 12cm from anal verge
* Clinical stage T2N+ or T3-4aNany,M0 Clinical staging should be estimated based on the combination of the following assessments: physical examination by the primary surgeon, CT scan of the chest/abdomen/pelvis, and a pelvic MRI with or without an endorectal ultrasound (ERUS)
* No evidence that tumor is adjacent to (defined as within 2 mm of) the mesorectal fascia on pre-operative MRI
* No tumor causing symptomatic bowel obstruction
* No distant metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0, 1
* White Blood Cell (WBC) ≥ 4,000/mm³
* Platelets ≥ 100,000/mm³
* Hemoglobin > 10.0 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 1.5 times ULN
* Creatinine ≤ 1.5 times ULN
* No co-morbid illnesses or other concurrent disease that, in the judgment of the clinician obtaining informed consent, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens

Exclusion Criteria:

* Pregnant or nursing
* Patient of child-bearing potential is not willing to employ adequate contraception
* Not willing to return to enrolling medical site for all study assessments
* With other invasive malignancy ≤ 5 years prior to registration; exceptions are colonic polyps, non-melanoma skin cancer, or carcinoma-in-situ of the cervix
* Chemotherapy within 5 years prior to registration (hormonal therapy is allowable if the disease-free interval is ≥ 5 years)
* Prior pelvic radiation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 663 (Actual)
Dates: Start 2014-08-13 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Local-regional failure-free survival | Up to 5 years
  the time interval between the date of randomization and the date of local or regional progression/relapse, or death, whichever occurred first.regional progression/relapse, or death, whichever occurred first.

SECONDARY OUTCOMES:
Disease free survival | Up to 5 years
  the time interval between the date of randomization and the date of the first cancer-related event, second cancer, or death from any cause, whichever occurred first.
Pathologic complete response and tumor regression grade | Up to 18 weeks
  Pathological response will be made based on assessment of the surgical specimen at the primary treatment site. This assessment is made in addition to the AJCC 7th edition summary staging. A pCR must include no gross or microscopic tumor identified anywhere within the surgical specimen. This must include:
  * No evidence of malignant cells in the primary tumor specimen
  * No lymph nodes that contain tumor. The definition of a non-pCR will include any surgical specimen that has any evidence of residual tumor manifest in the primary or regional lymph nodes. For patients who do not meet criteria for a pCR, the extent of response to preoperative therapy will be graded using the Tumor Regression Grade (TRG) schema that is included in the AJCC 7th edition. This was also used by Rodel in the pre/postoperative rectal cancer study and was subsequently adopted by the AJCC [Rodel (JCO 2005; 23:8688-8696)].
Pelvic R0 resection rate | Up to 18 weeks
  R0 resection: All gross disease has been removed, and microscopic examination reveals all surgical margins free of tumor.
Overall survival | Up to 5 years
  the time interval between the date of randomization to the date of death. If the patient has been alive, the time until the last follow-up is taken as the overall survival period.
Adverse event (AE) profiles | Up to 5 years
  The severity of AE and the laboratory findings were graded by the investigators according to Common Terminology Criteria for Adverse Events, version 4. All appropriate treatment areas should have access to a copy of the CTCAE version 4.0. A copy of the CTCAE version 4.0 can be downloaded from the CTEP web site: http://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm The maximum grade for each type of adverse events during neoadjuvant chemotherapy and chemoradiation therapy, and surgical complications will be recorded for each patient.
  Follow-up for patient safety should be done during the treatment period and 30 days after the end of the last cycle. The reason for the delay or interruption should be recorded on the CRF form.
Rate of receiving pre-operative or post-operative chemoradiation | Up to 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peirong Ding, MD, Ph D, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Mei WJ, Wang XZ, Li YF, Sun YM, Yang CK, Lin JZ, Wu ZG, Zhang R, Wang W, Li Y, Zhuang YZ, Lei J, Wan XB, Ren YK, Cheng Y, Li WL, Wang ZQ, Xu DB, Mo XW, Ju HX, Ye SW, Zhao JL, Zhang H, Gao YH, Zeng ZF, Xiao WW, Zhang XP, Zhang X, Xie E, Feng YF, Tang JH, Wu XJ, Chen G, Li LR, Lu ZH, Wan DS, Bei JX, Pan ZZ, Ding PR. Neoadjuvant Chemotherapy With CAPOX Versus Chemoradiation for Locally Advanced Rectal Cancer With Uninvolved Mesorectal Fascia (CONVERT): Initial Results of a Phase III Trial. Ann Surg. 2023 Apr 1;277(4):557-564. doi: 10.1097/SLA.0000000000005780. Epub 2022 Dec 20. PMID 36538627